CLINICAL TRIAL: NCT04544735
Title: Integrated Physical Therapy and Coping Skills Training for Improving Women's Sexual Function After Pelvic Radiation
Brief Title: Improving Women's Function After Pelvic Radiation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00105435
Record Dates: First submitted 2020-09-04; First posted 2020-09-10 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Sexual Dysfunction; Pelvic Floor Disorders; Gynecologic Cancer
Keywords: Pelvic radiation; Sexual side effects; Pelvic health physical therapy; Cancer survivors; Intimacy dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrated Physical Therapy and Coping Skills Training (Experimental): The proposed intervention will will integrate two key components: pelvic health PT interventions (i.e., vaginal dilators, Pelvic Floor Muscle Training) and coping skills training for managing symptoms and improving treatment adherence. The intervention aims to improve women's sexual function after pelvic radiation
  Interventions: Behavioral: Integrated Physical Therapy and Coping Skills Training

INTERVENTIONS:
Behavioral: Integrated Physical Therapy and Coping Skills Training — The proposed intervention will provide pelvic health physical therapy interventions including: education about vaginal moisturizers and lubricants, low back and hip assessment and instruction in accommodations (e.g., strategies for accommodating sexual position of choice), instruction in vulvar massage, instruction and facilitation of vaginal dilator use, and pelvic floor muscle training (PFMT) and exercises. Women will be given a set of vaginal dilators. Cognitive behavioral techniques that have been successfully used by physical therapists in prior intervention studies will be integrated into the PT intervention including breathing and relaxation techniques, guided imagery, systematic desensitization, cognitive restructuring techniques and coping thoughts, and problem solving

SUMMARY:
The purpose of the study is to develop and test an intervention combining physical therapy (PT) and coping skills training to improve women's sexual function after pelvic radiation.

DETAILED DESCRIPTION:
Pelvic radiation, which is a critical component in the treatment of many gynecologic, bladder, rectal and anal cancers, often results in devastating and long-lasting sexual side effects. Vaginal changes following pelvic radiation include adhesions, agglutination, fibrosis, dryness, atrophy, and stenosis. Pelvic radiation-related sexual problems are often undertreated, resulting in poor symptom management and reduced quality of life. Rehabilitation programs including pelvic floor muscle training (PFMT) and vaginal dilator exercises may help minimize post-radiation vaginal changes and related sexual problems, but use of these rehabilitation strategies is inconsistent and infrequent in routine clinical practice. For many women, engaging in these rehabilitation strategies can be difficult and adherence is low (e.g.,1% to 35% for dilator use). Barriers to engaging in PFMT and dilator exercises include lack of information, pain, embarrassment, fear, and reliving invasive treatments. There is a critical need for interventions to help women access and engage in rehabilitation following pelvic radiation treatment. We propose to develop and pilot test a novel physical therapist delivered intervention to improve women's sexual function after pelvic radiation that integrates pelvic health physical therapy interventions (i.e., vaginal dilators, PFMT) and cognitive-behavioral based coping skills training for managing symptoms and improving treatment adherence. Pelvic health physical therapy interventions have demonstrated effectiveness for treating pelvic pain and sexual pain disorders. Coping skills training interventions have demonstrated benefits for reducing symptoms and improving treatment engagement.This study includes two phases: intervention development and pilot testing. For intervention development (months 1-6), qualitative data obtained from patient and healthcare provider interviews will be used to develop and refine the integrated PT and coping skills training intervention. Using information obtained in qualitative interviews, we will develop the intervention. In pilot testing (months 7-12), we will pilot the developed intervention with women who were treated with pelvic radiation. : The specific aims of this study are to: 1) develop and refine an integrated PT and coping skills training intervention based on qualitative data from interviews with cancer survivors, oncology providers, and pelvic health physical therapists; 2) pilot the developed intervention to examine its feasibility and acceptability; and 3) examine the patterns of change and relationships among outcome variables including vaginal changes, pelvic floor function, sexual function and satisfaction, and use of rehabilitation exercises.

ELIGIBILITY:
Cancer Survivors participating in the Intervention Development Interviews

Inclusion Criteria:

* Diagnosis of non-metastatic gynecologic (cervical, endometrial, vaginal, vulvar), anal, rectal, or bladder cancer
* Completed pelvic radiation treatment within the last 5 years
* 18 years of age or older
* Able to speak/read English
* Able to give meaningful informed consent

Exclusion Criteria:

* Major untreated or uncontrolled mental illness (e.g., schizophrenia)
* Unable to provide informed consent

Medical Providers Participating in Intervention Development Interviews

Eligibility Criteria:

* Oncology providers (e.g., radiation, medical, and surgical oncologists; nurses; advanced practice professionals) who provide care to women who receive pelvic radiation for gynecologic, anal, rectal or bladder cancers.
* Physical therapists with specialized certification in pelvic health or women's health physical therapy who provide care to patients in the outpatient setting.

Cancer Survivor User Testers

Inclusion Criteria:

* Diagnosis of non-metastatic gynecologic (cervical, endometrial, vaginal, vulvar), anal, rectal, or bladder cancer
* Completed pelvic radiation treatment in the past 2 to 24 months
* 18 years of age or older
* Able to speak/read English
* Able to give meaningful informed consent

Exclusion Criteria:

* Major untreated or uncontrolled mental illness (e.g., schizophrenia)
* Unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Session Attendance | Following completion of the intervention, up to 12 months
  Treatment feasibility will be assessed by measuring the session attendance rate for each participant
Attkisson & Zwick's Client Satisfaction Questionnaire | 3 months post intervention
  18 item questionnaire to measure and assess consumer satisfaction with health and human services.

SECONDARY OUTCOMES:
Sexual Vaginal Changes Questionnaire | Baseline and 3 months post intervention
  27-item questionnaire to assess intimacy, sexual interest, sexual satisfaction, vaginal changes (lubrication, pain and bleeding) and sexual functioning
Australian Pelvic Floor Questionnaire | Baseline and 3 month post intervention
  42 item questionnaire to assesses all pelvic floor symptoms including bladder, bowel and sexual function and prolapse symptoms
PROMIS Sexual Function and Satisfaction Measure Full Profile (Female) | Baseline and 3 months post intervention
  27 item questionnaire to measure sexual function and satisfaction in female population with cancer in past 30 days
Generalized Anxiety Disorder Screener (GAD-7) | Baseline and 3 months post intervention
  7-item questionnaire to assess symptoms of anxiety over the past two weeks
Patient Health Questionnaire Depression Screener (PHQ-9) | Baseline and 3 months post intervention
  9-item questionnaire to asses depressive symptoms over the past two weeks
Adherence to Rehabilitation Strategies Scale | Baseline and 3 months post intervention
  3 item questionnaire to assess adherence to rehabilitation strategies such as vaginal dilators, moisturizers, pelvic floor muscle exercises.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Shelby, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No